CLINICAL TRIAL: NCT02371304
Title: Rectal Preserving Treatment for Early Rectal Cancer. A Multi-centred Randomised Trial of Radical Surgery Versus Adjuvant Chemoradiotherapy After Local Excision for Early Rectal Cancers
Acronym: TESAR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Jurriaan B. Tuynman, MD, PhD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL50364.029
Record Dates: First submitted 2015-02-18; First posted 2015-02-25 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Rectal Cancer
Keywords: Local therapy; Adjuvant chemoradiotherapy; Rectal preserving
MeSH Terms: conditions — Rectal Neoplasms | interventions — Chemoradiotherapy, Adjuvant; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Total Mesorectal Excision (Active Comparator): After local excision patients will receive additional TME surgery
  Interventions: Procedure: Additional TME surgery
- Adjuvant chemoradiotherapy (Experimental): After local excision. Patients will receive capecitabine 825 mg/m2 twice a day for 5 weeks only on weekdays. This will be combined with 1.8 Gy in 25 fractions with a limited dose only on the mesorectum
  Interventions: Radiation: Adjuvant chemoradiotherapy; Drug: capecitabine

INTERVENTIONS:
Radiation: Adjuvant chemoradiotherapy — Patients will receive capecitabine 825 mg/m2 twice a day for 5 weeks only on weekdays. This will be combined with 1.8 Gy in 25 fractions with a limited dose only on the mesorectum
  Arms: Adjuvant chemoradiotherapy
Procedure: Additional TME surgery
  Arms: Total Mesorectal Excision
Drug: capecitabine
  Arms: Adjuvant chemoradiotherapy

SUMMARY:
Current therapy for early colorectal cancer is radical Total Mesorectal Excision (TME). Colorectal surgical resections are accompanied with high morbidity of up to 33% and 90 days mortality of up to 9% in the fragile elderly patients as is seen in the results of the Dutch Surgical Colorectal Audit (DSCA) of 2013. Additionally, rectal cancer surgery is associated with substantial loss of health related quality of life due to defecation disorders, incontinence, sexual dysfunction and stoma related morbidity. These disadvantages are acceptable when radical surgery is the only option for cure. Advances in technology enabled the development of local excision of early rectal cancer with precise endoluminal microsurgery or local endoscopic excision resulting in a significant decrease in short- and long term morbidity. However current evidence is of inadequate quality to conclude on the oncologic safety of local treatment for early rectal cancer. Imaging can predict outcome and tailors treatment in more advanced cancer but fails in early cancer. Pathological assessment of the excised tumor tissue provides the optimal information on tumor stage, tumor characteristics and tumor differentiation, thereby it enables to predict the risk of recurrence after local treatment alone. For early rectal cancers, with a low risk on recurrence based on favourable tumor characteristics local excision is seen as safe and these patients do not require an additional treatment. However, for patients with early rectal cancer with a higher risk on recurrence based on tumor characteristics there is no consensus on the additional treatment after local excision. According to the National guideline these patients receive a TME procedure. However, for this subgroup of patients local treatment followed by chemoradiotherapy might also be oncological safe. Current evidence is of inadequate quality to be conclusive. For this subgroup of patients with early rectal cancer with high risk tumorcharacteristics the TESAR trial is designed, in which patiens will be randomised after local endoluminal excision between an additional TME-procedure (standard) and adjuvant chemoradiotherapy. Primary endpoint of the study will be local recurrence at 3 three year follow-up.

ELIGIBILITY:
Inclusion criteria:

1. Patient has had an endoluminal local excision (by TEM, TAMIS, TSPM, EMR/ESD or polypectomy) of an early rectal cancer without carcinoma in the resection plane.
2. Patients with carcinoma in the resection plane or in case of unreliable resection planes (EMR/ESD) no macroscopic residual tumour confirmed by endoscopy are eligible for randomisation.
3. Only lesions for which TME surgery is indicated can be included (if a partial mesorectal excision (PME) is indicated the patient should be excluded).
4. Pathological confirmation of the rectal adenocarcinoma fulfilling the following criteria: T1 with size 3-5 cm of carcinoma or pT1, maximum size of carcinoma of 3 cm, with at least poor differentiation, Haggit 4 and/or sm3, lymphatic and/or venous invasion.
5. Pathological confirmation of the rectal adenocarcinoma fulfilling the following criteria: pT2, maximum size of carcinoma of 3 cm, well/moderate differentiated and without lymphatic or venous invasion.
6. Complete colonoscopy, without synchronous colorectal cancer.
7. cN0 stage based on pelvic MRI; lymph nodes smaller than 10 mm will be considered as benign, independent of morphologic features. Staging done within 6 weeks before randomisation.
8. Adequate distant staging (X-thorax or CT-thorax and CT-abdomen) without signs of distant metastasis (cM0).
9. Male or female, Age > 18 years.
10. Life expectancy of at least 12 months.
11. Medically fit (WHO 0-2) to undergo radical surgery and/or radiation.
12. No contraindications to chemotherapy, including adequate blood counts;

    * white blood count >= 4.0 x 10 9/l
    * platelet count >=100 x 109/l
    * clinical acceptable haemoglobin levels
    * bilirubin < 35 umol/l
    * creatinine levels indicating renal clearance of >=50 ml/min
13. The patient is willing and able to comply with the protocol for the duration of the study, and scheduled follow-up visits and examinations.
14. Written (signed and dated) informed consent and be capable of co-operating with protocol.

Exclusion Criteria:

1. Incomplete or inconclusive resection margin with macroscopic residual tumour.
2. T1 tumour with carcinoma < 3 cm, moderate/well differentiated, without sm3, venous or lymphatic invasion.
3. T1 tumour with carcinoma of >5 cm and T2 tumour with carcinoma of > 3 cm.
4. Presence of metastatic disease or recurrent rectal tumour.
5. Previous pelvic radiation.
6. Treatment with any other investigational agent, or participation in another clinical trial within 28 days prior to enrolment.
7. Concomitant malignancies, except for adequately treated basocellular carcinoma of the skin or in situ carcinoma of the cervix uteri. Subjects with prior malignancies must be disease-free for at least 5 years.
8. Pregnancy, breast-feeding or fertile women without active birth control.
9. Clinically significant (i.e. active) cardiovascular disease for example cerebro vascular accidents (<6 months prior to randomization), myocardial infarction (<6 months prior to randomization), unstable angina, New York Heart Association (NYHA) grade II or higher, congestive heart failure, serious cardiac arrhythmia requiring medication.
10. Patients who are known to be serologically positive for Hepatitis B, Hepatitis C or HIV.
11. History of severe and unexpected reactions to fluoropyrimidine therapy.
12. Hypersensitivity to capecitabine.
13. Patients with severe hepatic impairment.
14. Medical or psychiatric conditions that compromise the patient's ability to give informed consent.
15. Patients known with dihydropyrimidine dehydrogenase deficiency
16. Any contra-indications to undergo MRI imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2015-10; Primary Completion 2022-06 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence free at 3 year follow-up | 3 year

SECONDARY OUTCOMES:
Treatment related morbidity | 1,3 and 5 year follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Borstlap WA, Tanis PJ, Koedam TW, Marijnen CA, Cunningham C, Dekker E, van Leerdam ME, Meijer G, van Grieken N, Nagtegaal ID, Punt CJ, Dijkgraaf MG, De Wilt JH, Beets G, de Graaf EJ, van Geloven AA, Gerhards MF, van Westreenen HL, van de Ven AW, van Duijvendijk P, de Hingh IH, Leijtens JW, Sietses C, Spillenaar-Bilgen EJ, Vuylsteke RJ, Hoff C, Burger JW, van Grevenstein WM, Pronk A, Bosker RJ, Prins H, Smits AB, Bruin S, Zimmerman DD, Stassen LP, Dunker MS, Westerterp M, Coene PP, Stoot J, Bemelman WA, Tuynman JB. A multi-centred randomised trial of radical surgery versus adjuvant chemoradiotherapy after local excision for early rectal cancer. BMC Cancer. 2016 Jul 21;16:513. doi: 10.1186/s12885-016-2557-x. PMID 27439975